CLINICAL TRIAL: NCT02519452
Title: An Open-label, Multicenter, Dose Escalation Phase 1b Study to Assess the Safety and Pharmacokinetics of Subcutaneous Delivery of Daratumumab With the Addition of Recombinant Human Hyaluronidase (rHuPH20) for the Treatment of Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Daratumumab With the Addition of Recombinant Human Hyaluronidase (rHuPH20) for the Treatment of Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR107838; 2015-001210-94 (EudraCT Number); 54767414MMY1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Daratumumab (JNJ-54767414); Recombinant Human Hyaluronidase
MeSH Terms: conditions — Multiple Myeloma | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (5):
- Part 1: Cohort 1 (Experimental): Participants will receive 1200 mg (daratumumab 1200 milligram (mg) with Recombinant Human Hyaluronidase [rHuPH20] 30,000 U) via mixing immediately before Subcutaneous (SC) infusion once weekly in Cycles 1 (each cycle is 28 days) and 2, every 2 weeks in Cycles 3-6, and then every 4 weeks in subsequent cycles until disease progression.
  Interventions: Drug: Daratumumab Subcutaneous (SC) Administration; Drug: Recombinant Human Hyaluronidase [rHuPH20]) SC Administration
- Part 1: Cohort 2 (Experimental): Participants will receive 1800 mg (daratumumab 1800 milligram (mg) with Recombinant Human Hyaluronidase [rHuPH20] 45,000 U) via mixing immediately before SC infusion once weekly in Cycles 1 and 2, every 2 weeks in Cycles 3-6, and then every 4 weeks in subsequent cycles until disease progression.
  Interventions: Drug: Daratumumab Subcutaneous (SC) Administration; Drug: Recombinant Human Hyaluronidase [rHuPH20]) SC Administration
- Part 1: Cohort 3 (Experimental): Participants will receive mixture of daratumumab and rHuPH20 prepared immediately before administration via Subcutaneous (SC) delivery at a dose which will be decided by Study Evaluation Team (SET) once weekly by SC infusion in Cycles 1 and 2, every 2 weeks in Cycles 3-6, and then every 4 weeks in subsequent cycles until disease progression. Also up to three additional optional cohorts (Cohorts 3b, 3c, and 3d) may be enrolled to repeat a dose level of daratumumab.
  Interventions: Drug: Daratumumab Subcutaneous (SC) Administration; Drug: Recombinant Human Hyaluronidase [rHuPH20]) SC Administration
- Part 2: Cohort 4 (Experimental): Participants will receive 1800 mg co-formulated daratumumab and rHuPH20 preparation initially administered by SC injection once weekly in Cycles 1 and 2, every 2 weeks in Cycles 3-6, and then every 4 weeks in subsequent cycles. The dose level and schedule for any additional cohorts would be selected based on the daratumumab pharmacokinetic profile and safety profile (reviewed by the SET) that will be observed in Cohort 4.
  Interventions: Drug: Daratumumab Subcutaneous (SC) Administration; Drug: Recombinant Human Hyaluronidase [rHuPH20]) SC Administration
- Part 3: Dara-CF 1800 mg (Experimental): Participants will receive co-formulated daratumumab 1800 mg and rHuPH20 preparation (Dara-CF) initially administered by SC injection once weekly in Cycles 1 and 2, every 2 weeks in Cycles 3-6, and then every 4 weeks in subsequent cycles.
  Interventions: Drug: Daratumumab Subcutaneous (SC) Administration; Drug: Recombinant Human Hyaluronidase [rHuPH20]) SC Administration

INTERVENTIONS:
Drug: Daratumumab Subcutaneous (SC) Administration — Participants will receive Daratumumab mixed with rHuPH20 in part 1 and co-formulated with rHuPH20 in part 2 and part 3 administered via SC administration once weekly in Cycles 1 (each cycle is 28 days) and 2, every 2 weeks in Cycles 3-6, and every 4 weeks in subsequent cycles.
Drug: Recombinant Human Hyaluronidase [rHuPH20]) SC Administration — Participants will receive Recombinant Human Hyaluronidase [rHuPH20]) mixed with Daratumumab in part 1 and co-formulated with Daratumumab in part 2 and part 3 administered as SC administration once weekly in Cycles 1 (each cycle is 28 days) and 2, every 2 weeks in Cycles 3-6, and every 4 weeks in subsequent cycles.

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics and safety from the mixture of daratumumab and rHuPH20 prepared immediately before administration via Subcutaneous (SC) delivery (Part 1) and CF (co-formulated daratumumab and rHuPH20 preparation) administration via SC delivery of daratumumab (Part 2) and to evaluate the safety of Dara-CF 1800 milligram (mg) SC delivery without pre-dose and post-dose corticosteroids (Part 3).

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known), multicenter, 3-part, Phase 1b dose escalation/expansion study to evaluate the safety, pharmacokinetics (study of what the body does to a drug), and antitumor activity of SC delivery of daratumumab to participant with relapsed or refractory multiple myeloma. Up to approximately 53 participants in part 1, 80 participants in part 2 and 15 participants per corticosteroid tapering cohort (up to approximately 30 participants total) in Part 3 will be enrolled. The purpose of Part 1 is to select an appropriate SC therapeutic dose for the mixture of daratumumab with rHuPH20 based on safety and pharmacokinetics. This dose, selected from part 1 will be the initial dose for the co-formulated daratumumab and rHuPH20 preparation to be evaluated in Part 2. The purpose of Part 2 is to evaluate the SC delivery of CF and confirm the dose level selected from Part 1 based on the pharmacokinetics, safety, and antitumor activity. The purpose of Part 3 is to evaluate the safety of Dara-CF 1800 mg SC delivery without pre-dose and post-dose corticosteroids. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants proven to have multiple myeloma (MM) diagnosis according to the International Myeloma Working Group (IMWG) diagnostic criteria
* Measurable disease as defined by any of the following: (a) immunoglobulin (Ig) G myeloma (serum monoclonal paraprotein [M-protein] level >=1.0 gram/deciliter [g/dL] or urine M-protein level greater than or equal to (>=) 200 milligram[mg]/24 hours[hrs]; or (b) IgA, IgD, or IgE multiple myeloma (serum M-protein level >= 0.5 g/dL or urine M-protein level >= 200 mg/24 hrs); or (c) light chain multiple myeloma (serum immunoglobulin free light chain >=10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio)
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Pretreatment clinical laboratory values must meet protocol-defined parameters during the Screening phase
* Man, who is sexually active with a woman of child-bearing potential and has not had a vasectomy, must agree to use a barrier method of birth control example (eg), either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the final dose of study drug
* Relapsed or refractory disease. Relapse is defined as progression of disease after an initial response to previous treatment, more than 60 days after cessation of treatment. Refractory disease is defined as less than (<) 25 percent (%) reduction in M-protein or progression of disease during treatment or within 60 days after cessation of treatment
* Prior treatment with less than or equal to (>=) 2 treatment lines of anti-myeloma therapy. Prior lines of therapy must include a proteasome inhibitor (PI) (eg, bortezomib, carfilzomib) and an immunomodulatory drug (IMiD) (example, thalidomide, lenalidomide, pomalidomide) in any order during the course of treatment. Each prior line of therapy may consist of one or more agents and may include induction, hematopoietic stem cell transplantation, and/or maintenance therapy. Radiotherapy, bisphosphonates, or a single short course of steroids is not considered a prior line of therapy

Exclusion Criteria:

* Participant has received daratumumab or other anti-cluster of differentiation 38 (anti-CD38) therapies previously
* Participant has received anti-myeloma treatment within 2 weeks before Cycle 1 Day 1
* Participant has previously received an allogenic stem cell transplant; or participant has received autologous stem cell transplantation (ASCT) within 12 weeks before Cycle 1 Day 1
* Participant has a history of malignancy (other than multiple myeloma) within 5 years before Cycle 1 Day 1 (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* Participant is exhibiting clinical signs of meningeal involvement of multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Serum Trough Concentrations (Ctrough) of Daratumumab | Up to cycle 3 (each cycle 28 days) Day 1
  Ctrough: the concentration prior to study drug administration.
Part 1, 2 and 3: Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (30 days after last dose administration) (Approximately up to 3.4 years)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Part 1, 2 and 3: Serum Concentration of Daratumumab and Recombinant Human Hyaluronidase (rHuPH20) (Plasma) Antibodies | Approximately 2 years
  Serum levels of antibodies to Daratumumab and rHuPH20 for evaluation of potential immunogenicity.
Part 1, 2 and 3: Percentage of Participants with Complete Response (CR) | Approximately 2 years
  CR is Defined as the proportion of Participants achieving CR (including sCR) according to the International Myeloma Working Group (IMWG) criteria.
Part 1, 2 and 3: Percentage of Participants With Overall Response Rate (ORR) | Approximately 2 years
  Overall response rate is defined as the percentage of participants who achieve complete response, stringent complete response (sCR), partial response or very good partial response (VGPR) according to the International Myeloma Working Group criteria, during or after study treatment.
Part 1, 2 and 3: Duration of Response (DR) | Approximately 2 years
  The DR is time from date of initial documentation of response (PR or better) to date of first documented PD, as defined by IMWG criteria.
Part 1, 2 and 3: Time to Response | Approximately 2 years
  Time to response is defined as the time from the date of first dose of study treatment to the date of the first documentation of observed response (CR or PR or better than PR)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (12):
- United States (4):
  - Atlanta, Georgia
  - New York, New York
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
- Vejle, Denmark
- France (2):
  - Nantes
  - Tours
- Amsterdam, Netherlands
- Spain (3):
  - Badalona
  - Pamplona
  - Salamanca
- Stockholm, Sweden

REFERENCES:
- [Derived] Li X, Dosne AG, Perez Ruixo C, Perez Ruixo JJ. Pharmacodynamic-Mediated Drug Disposition (PDMDD) Model of Daratumumab Monotherapy in Patients with Multiple Myeloma. Clin Pharmacokinet. 2023 May;62(5):761-777. doi: 10.1007/s40262-023-01232-8. Epub 2023 Apr 6. PMID 37022569
- [Derived] Nahi H, Usmani SZ, Mateos MV, van de Donk NWCJ, Oriol A, Plesner T, Bandyopadhyay N, Hellemans P, Tromp B, Nnane I, Zemlickis D, Chari A, Moreau P. Corticosteroid tapering is a safe approach in patients with relapsed or refractory multiple myeloma receiving subcutaneous daratumumab: part 3 of the open-label, multicenter, phase 1b PAVO study. Leuk Lymphoma. 2023 Feb;64(2):468-472. doi: 10.1080/10428194.2022.2148221. Epub 2023 Jan 2. No abstract available. PMID 36593729
- [Derived] Usmani SZ, Nahi H, Mateos MV, van de Donk NWCJ, Chari A, Kaufman JL, Moreau P, Oriol A, Plesner T, Benboubker L, Hellemans P, Masterson T, Clemens PL, Luo M, Liu K, San-Miguel J. Subcutaneous delivery of daratumumab in relapsed or refractory multiple myeloma. Blood. 2019 Aug 22;134(8):668-677. doi: 10.1182/blood.2019000667. Epub 2019 Jul 3. PMID 31270103